CLINICAL TRIAL: NCT05086146
Title: Prognostic Impact of Cardiac Imaging During Suspected Immune Checkpoint Inhibitor Myocarditis
Acronym: IMMUNOIMAGING
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-63; 2020-A03384-35 (Other: IDRCB)
Record Dates: First submitted 2021-09-23; First posted 2021-10-20 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Myocarditis
MeSH Terms: conditions — Myocarditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
It consists of evaluating the advantage of routine detection of phIGFBP-1 to reduce the total duration of hospitalization for patients with a risk of preterm labor before 32 weeks of gestation without increasing the number of preterm labour.

DETAILED DESCRIPTION:
Patient with a risk of preterm labor (ultrasound cervical length < 25 mm +/- described or recorded uterine contractions) before 32 weeks of gestation will be hospitalized to receive tocolytic drugs and antenatal corticosteroid therapy according to the investigators gold standard protocol. After 48 hours, the participants will be assessed by examination, external tocodynamometry and the measure of cervical length by ultrasound. Stabilized patients will be included and randomized into 2 groups of 210 patients each. The first group "A" will benefit from the standard protocol (extended hospitalization of 2 or 4 days according to the clinical and ultrasound assessment); whereas the second group, "B", will have the benefit of the detection of phIGFBP-1.If the result proves negative, patients could be discharged early at day 2. In the case of a positive result, patients will follow the standard procedure because of the low positive predictive value of the test. The main outcome is the total duration of hospitalization.

ELIGIBILITY:
Inclusion Criteria:

All patients affiliated to the French social security system will be eligible, after signing a consent form, and presenting the following criteria

* Introduction within the last 3 months of at least one of the following ICIs: nivolumab, pembrolizumab, cemiplimab, avelumab, atezolizumab, ipilimumab, tremelimumab, durvalumab.
* Suspicion of myocarditis defined by the presence of at least one of the following criteria adapted from the European Society of Cardiology guidelines:

  * Symptomatic patients (chest pain, dyspnea, palpitations, syncope/lipothymia) within 7 days of ICI administration
  * New ECG abnormality (ST-segment elevation, ST-segment undershift, arrhythmia, conductive disturbances, T-wave inversion)
  * Elevation of troponin above the 99th percentile of the laboratory reference value or, if troponin is already elevated before treatment, an increase of more than 30% of the baseline value
  * Recent LVEF decline or recent LV contraction abnormality on a TTE
* Patient has given no objection

Translated with www.DeepL.com/Translator (free version)

Exclusion Criteria:

* Age <18 years
* Major under guardianship or curatorship
* Pregnant or breastfeeding women
* Patient not covered by a social security plan
* Hemodynamic or rhythmic instability
* Estimation of glomerular filtration rate by the MDRD formula <30ml/min/1.73m2
* Implantable equipment that does not allow for cMRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients with suspected myocarditis on ICIs.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-08-10 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence rate of the composite end point | 6-month
  including cardiovascular death, acute heart failure, cardiogenic shock, cardiac arrest, sustained ventricular tachycardia, ventricular fibrillation, 2nd-degree (except Mobitz 1) or 3rd-degree atrioventricular block.

SECONDARY OUTCOMES:
Cumulative incidence rate of all-cause death | 6-month

CONTACTS AND LOCATIONS:
Overall Officials: François CREMIEUX, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- assistance publique hôpitaux de Marseille, Marseille, France